CLINICAL TRIAL: NCT01277250
Title: Web-based Smoking Cessation Intervention: Transition From Inpatient to Outpatient
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1U01DA031515 (NIH)
Record Dates: First submitted 2011-01-12; First posted 2011-01-14 (Estimated); Last update posted 2015-06-19 (Estimated); Status verified 2015-06

CONDITIONS: Cigarette Smoking; Home Access to Internet and Email; Cognitively and Physically Able to Participate; English Speaking and Reading
Keywords: Hospitalized adults; Tobacco users; Smokers; Smoking cessation; Web-based; Transition coach
MeSH Terms: conditions — Cigarette Smoking; Tobacco Use; Smoking Cessation | interventions — Behavior Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Usual Care (Other): Standard smoking cessation information provided to all hospitalized patients as part of discharge packet.
  Interventions: Behavioral: Web-based smoking cessation program
- Smoking Cessation Program (Experimental): Web-based program tailored to patients who smoke and are hospitalized. Program is tailored to participant's specific hospital experience and other characteristics. E-messages, social support and a "transition coach" are provided to each participant in this condition.
  Interventions: Behavioral: Web-based smoking cessation program

INTERVENTIONS:
Behavioral: Web-based smoking cessation program — Web-based smoking cessation program that includes a "transition coach" to hospitalized patients who will assist them in quitting as they are discharged from the hospital. Intervention arm participants will have access to a tailored web-based intervention that will include e-messages and activities that are tailored to their recent hospital stay.
  Other Names: Tobacco Treatment; Behavioral Counseling; Computer-Assisted Treatment

SUMMARY:
This project, "Web-based Smoking Cessation Intervention: transition from inpatient to outpatient," addresses smoking among hospitalized patients, whose rates are higher than among the general population. Hospitalization offers a unique opportunity to intervene, as it requires temporary abstinence and patients are focused on health concerns. Hypotheses: A tailored web-based and e-message smoking cessation program for current smokers that, upon hospital discharge, transitions the patient to continue a quit attempt when home will be effective. Further, the investigators hypothesize that this approach will be cost-effective. Specific Aims: 1. To test the effectiveness of a web-based smoking cessation intervention. 2. To determine the cost-effectiveness of this approach. Research Design - Methods: A randomized two-arm follow-up design will be used to test the effectiveness of an evidence- and theoretically-based smoking cessation program designed for post-hospitalization. Patients randomized to this arm will be contacted by hospital staff, trained as 'transition coaches,' to engage in Decide2Quit, an interactive web-based program that offers personalized and tailored messages, e-group support, and text messages promoting tobacco abstinence. All hospitalized patients will receive standardized smoking cessation materials. As well, physicians can order nicotine replacement therapy via the hospital's electronic order system. The investigators primary outcome is biologically confirmed and self-reported tobacco abstinence at 6 months follow-up; the investigators will also assess self-reported quit rates at 3 and 12 months and variables hypothesized to predict quit success. We will measure health care utilization and quality of life to allow testing the cost-effectiveness of this program conducted from the perspective of a hospital, health care payers, patients and society. Significance of results: At study completion the investigators will know whether imbedding smoking cessation into usual hospital care, with minimal hospital-staff burden, and an interactive web-based tailored intervention program is an effective way to reduce smoking rates among hospitalized patients, and if it is cost-effective. This program will be an "off the shelf approach that could be disseminated easily.

ELIGIBILITY:
Inclusion Criteria:

* 19 years of age or older
* Current smoker (at least one puff in the last 30 days)
* Regular (at least weekly) email/internet access
* Can read and speak English
* Can communicate well enough to provide meaningful responses to the screening questions and informed consent
* Well enough to participate (provide meaningful responses to the screening questions and informed consent)
* On standard or contact isolation only
* Cognitively able to participate (to provide meaningful responses to the screening questions and informed consent)
* Does not have another household member participating in this study

Exclusion Criteria:

* Under age 19
* Non-smoker
* Cannot read and speak English
* No email/internet access
* Cannot communicate well enough to provide meaningful responses to the screening questions and informed consent
* Too ill to participate (provide meaningful responses to the screening questions and informed consent)
* On isolation precautions other than standard or contact
* Cognitively unable to participate (to provide meaningful responses to the screening questions and informed consent)
* Has another household member participating in this study

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1548 (Actual)
Dates: Start 2011-07; Primary Completion 2014-09 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Smoking abstinence | 6 months
  Biochemically-verified (cotinine) and self-reported tobacco abstinence

SECONDARY OUTCOMES:
Smoking abstinence | 3 and 12 months
  self-reported tobacco abstinence

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen F Harrington, PhD, MPH, Principal Investigator — The University of Alabama at Birmingham
Locations (1):
- The University of Alabama at Birmingham - Lung Health Center, Birmingham, Alabama, United States

REFERENCES:
- [Background] Centers for Disease Control and Prevention (CDC). Cigarette smoking among adults--United States, 2007. MMWR Morb Mortal Wkly Rep. 2008 Nov 14;57(45):1221-6. PMID 19008790
- [Background] Centers for Disease Control and Prevention (CDC). State-specific prevalence and trends in adult cigarette smoking--United States, 1998-2007. MMWR Morb Mortal Wkly Rep. 2009 Mar 13;58(9):221-6. PMID 19282813
- [Background] Boyle RG, Solberg LI, Asche SE, Maciosek MV, Boucher JL, Pronk NP. Proactive recruitment of health plan smokers into telephone counseling. Nicotine Tob Res. 2007 May;9(5):581-9. doi: 10.1080/14622200701243201. PMID 17454714
- [Background] Rigotti NA, Munafo MR, Stead LF. Smoking cessation interventions for hospitalized smokers: a systematic review. Arch Intern Med. 2008 Oct 13;168(18):1950-60. doi: 10.1001/archinte.168.18.1950. PMID 18852395
- [Background] Mohiuddin SM, Mooss AN, Hunter CB, Grollmes TL, Cloutier DA, Hilleman DE. Intensive smoking cessation intervention reduces mortality in high-risk smokers with cardiovascular disease. Chest. 2007 Feb;131(2):446-52. doi: 10.1378/chest.06-1587. PMID 17296646
- [Background] Katz A, Goldberg D, Smith J, Trick WE. Tobacco, alcohol, and drug use among hospital patients: concurrent use and willingness to change. J Hosp Med. 2008 Sep;3(5):369-75. doi: 10.1002/jhm.358. PMID 18951399
- [Background] Division of Chronic Disease Prevention and Control. Illinois Department of Public Health Tobacco Burden in Illinois 2005. Springfield, IL: Illinois Department of Public Health; 2005.
- [Background] Reid RD, Mullen KA, Slovinec D'Angelo ME, Aitken DA, Papadakis S, Haley PM, McLaughlin CA, Pipe AL. Smoking cessation for hospitalized smokers: an evaluation of the "Ottawa Model". Nicotine Tob Res. 2010 Jan;12(1):11-8. doi: 10.1093/ntr/ntp165. Epub 2009 Nov 10. PMID 19903737
- [Background] Shields M. Smoking-prevalence, bans and exposure to second-hand smoke. Health Rep. 2007 Aug;18(3):67-85. No abstract available. PMID 17892252
- [Background] Benowitz NL, Schultz KE, Haller CA, Wu AH, Dains KM, Jacob P 3rd. Prevalence of smoking assessed biochemically in an urban public hospital: a rationale for routine cotinine screening. Am J Epidemiol. 2009 Oct 1;170(7):885-91. doi: 10.1093/aje/kwp215. Epub 2009 Aug 27. PMID 19713287
- [Background] California Department of Health Services, Section TC. Adult Smoking Prevalence. http.//www.dhs.ca.gov/tobacco. Accessed January 6, 2010.
- [Background] The Joint Commission. Comprehensive Accreditation Manual for Hospitals. http://www.jcrinc.com/Joint-Commission-Requirements/Hospitals/. Accessed January 13, 2010.
- [Background] Freund M, Campbell E, Paul C, Sakrouge R, Lecathelinais C, Knight J, Wiggers J, Walsh RA, Jones T, Girgis A, Nagle A. Increasing hospital-wide delivery of smoking cessation care for nicotine-dependent in-patients: a multi-strategic intervention trial. Addiction. 2009 May;104(5):839-49. doi: 10.1111/j.1360-0443.2009.02520.x. Epub 2009 Mar 13. PMID 19344446
- [Background] Center for Medicare and Medicaid Services. Electronic Medical Records. http://search.cms.hhs.gov/search?q=electronic+medical+record&site=cms_collection&output=xml_no_dtd&client=cms_frontend&proxystylesheet=cms_frontend&oe=UTF-8&ie=UTF-8&ip=10.10.4.252&access=p&sort=date%3AD%3AL%3Ad1&entqr=0&ud=1&start=10. Accessed January 12, 2010.
- [Background] CDC. Tobacco-Related Costs and Expenditure in the United States. http://www.cdc.gov/tobacco/data_statistics/fact_sheets/fast_facts/index.htm. Accessed January 13, 2010.
- [Background] Glantz SA. Meta-analysis of the effects of smokefree laws on acute myocardial infarction: an update. Prev Med. 2008 Oct;47(4):452-3. doi: 10.1016/j.ypmed.2008.06.007. Epub 2008 Jun 18. No abstract available. PMID 18602944
- [Background] Centers for Disease Control and Prevention (CDC). Reduced hospitalizations for acute myocardial infarction after implementation of a smoke-free ordinance--City of Pueblo, Colorado, 2002-2006. MMWR Morb Mortal Wkly Rep. 2009 Jan 2;57(51):1373-7. PMID 19116606
- [Background] Pell JP, Haw S, Cobbe S, Newby DE, Pell AC, Fischbacher C, McConnachie A, Pringle S, Murdoch D, Dunn F, Oldroyd K, Macintyre P, O'Rourke B, Borland W. Smoke-free legislation and hospitalizations for acute coronary syndrome. N Engl J Med. 2008 Jul 31;359(5):482-91. doi: 10.1056/NEJMsa0706740. PMID 18669427
- [Background] Rigotti NA, Munafo MR, Murphy MF, Stead LF. Interventions for smoking cessation in hospitalised patients. Cochrane Database Syst Rev. 2003;(1):CD001837. doi: 10.1002/14651858.CD001837. PMID 12535418
- [Background] Tanni SE, Iritsu NI, Tani M, de Camargo PA, Sampaio MG, Godoy I, Godoy I. Risk perceptions and behavior among hospitalized patients with smoking-related diseases. Prev Chronic Dis. 2009 Oct;6(4):A138. Epub 2009 Sep 15. No abstract available. PMID 19755014
- [Background] Prochazka AV, Palisoc A. What is the best intervention to help hospitalized patients quit smoking? The Hospitalist. 2008(June 2008).
- [Background] Committee on Quality of Health Care in America IoM. Crossing the Quality Chasm. Washington, DC: National Academy Press; 2001.
- [Background] Personal Health Working Group. Connecting for Health. New York, NY: Markle Foundation, (www.connectingforhealth.org); 2006.
- [Background] Pagliari C, Detmer D, Singleton P. Potential of electronic personal health records. BMJ. 2007 Aug 18;335(7615):330-3. doi: 10.1136/bmj.39279.482963.AD. PMID 17703042
- [Background] National Research Council (US) Committee on Enhancing the Internet for Health Applications: Technical Requirements and Implementation Strategies. Networking Health: Prescriptions for the Internet. Washington (DC): National Academies Press (US); 2000. Available from http://www.ncbi.nlm.nih.gov/books/NBK44718/ PMID 20669497
- [Background] American Health Information Management Association; American Medical Informatics Association. The value of personal health records. A joint position statement for consumers of healthcare by the American Health Information Management Association and the American Medical Informatics Association. J AHIMA. 2007 Apr;78(4):22, 24. No abstract available. PMID 17455841
- [Background] Tang PC, Ash JS, Bates DW, Overhage JM, Sands DZ. Personal health records: definitions, benefits, and strategies for overcoming barriers to adoption. J Am Med Inform Assoc. 2006 Mar-Apr;13(2):121-6. doi: 10.1197/jamia.M2025. Epub 2005 Dec 15. PMID 16357345
- [Background] Anderson JG, Rainey MR, Eysenbach G. The impact of CyberHealthcare on the physician-patient relationship. J Med Syst. 2003 Feb;27(1):67-84. doi: 10.1023/a:1021061229743. PMID 12617199
- [Background] Liederman EM, Lee JC, Baquero VH, Seites PG. The impact of patient-physician Web messaging on provider productivity. J Healthc Inf Manag. 2005 Spring;19(2):81-6. PMID 15869217
- [Background] Liederman EM, Lee JC, Baquero VH, Seites PG. Patient-physician web messaging. The impact on message volume and satisfaction. J Gen Intern Med. 2005 Jan;20(1):52-7. doi: 10.1111/j.1525-1497.2005.40009.x. PMID 15693928
- [Background] Liederman EM, Morefield CS. Web messaging: a new tool for patient-physician communication. J Am Med Inform Assoc. 2003 May-Jun;10(3):260-70. doi: 10.1197/jamia.M1259. Epub 2003 Jan 28. PMID 12626378
- [Background] eRisk Guidelines: ERisk Working Group for Healthcare http://www.medem.com/phy/phy_eriskguidelines.cfm. 2005.
- [Background] Hobbs J, Wald J, Jagannath YS, Kittler A, Pizziferri L, Volk LA, Middleton B, Bates DW. Opportunities to enhance patient and physician e-mail contact. Int J Med Inform. 2003 Apr;70(1):1-9. doi: 10.1016/s1386-5056(03)00007-8. PMID 12706177
- [Background] Japuntich SJ, Zehner ME, Smith SS, Jorenby DE, Valdez JA, Fiore MC, Baker TB, Gustafson DH. Smoking cessation via the internet: a randomized clinical trial of an internet intervention as adjuvant treatment in a smoking cessation intervention. Nicotine Tob Res. 2006 Dec;8 Suppl 1:S59-67. doi: 10.1080/14622200601047900. PMID 17491172
- [Background] Myung SK, McDonnell DD, Kazinets G, Seo HG, Moskowitz JM. Effects of Web- and computer-based smoking cessation programs: meta-analysis of randomized controlled trials. Arch Intern Med. 2009 May 25;169(10):929-37. doi: 10.1001/archinternmed.2009.109. PMID 19468084
- [Background] Shahab L, McEwen A. Online support for smoking cessation: a systematic review of the literature. Addiction. 2009 Nov;104(11):1792-804. doi: 10.1111/j.1360-0443.2009.02710.x. PMID 19832783
- [Background] Bock BC, Graham AL, Whiteley JA, Stoddard JL. A review of web-assisted tobacco interventions (WATIs). J Med Internet Res. 2008 Nov 6;10(5):e39. doi: 10.2196/jmir.989. PMID 19000979
- [Background] Kushniruk A, Patel V, Cimino JJ, Barrows RA. Cognitive evaluation of the user interface and vocabulary of an outpatient information system. Proc AMIA Annu Fall Symp. 1996:22-6. PMID 8947620
- [Background] Nagle AL, Hensley MJ, Schofield MJ, Koschel AJ. A randomised controlled trial to evaluate the efficacy of a nurse-provided intervention for hospitalised smokers. Aust N Z J Public Health. 2005 Jun;29(3):285-91. doi: 10.1111/j.1467-842x.2005.tb00770.x. PMID 15991780
- [Background] Lancaster T, Silagy C, Fowler G. Training health professionals in smoking cessation. Cochrane Database Syst Rev. 2000;(3):CD000214. doi: 10.1002/14651858.CD000214. PMID 10908465
- [Background] Grimshaw GM, Stanton A. Tobacco cessation interventions for young people. Cochrane Database Syst Rev. 2006 Oct 18;(4):CD003289. doi: 10.1002/14651858.CD003289.pub4. PMID 17054164
- [Background] Dijkstra A, Vonk JM, Jongepier H, Koppelman GH, Schouten JP, ten Hacken NH, Timens W, Postma DS. Lung function decline in asthma: association with inhaled corticosteroids, smoking and sex. Thorax. 2006 Feb;61(2):105-10. doi: 10.1136/thx.2004.039271. Epub 2005 Nov 24. PMID 16308336
- [Background] Bandura A. Social Foundations of Thought and Action. Englewood Cliffs, N.J.: Prentice-Hall; 1986.
- [Background] Fiore MC, Jaen CR, Baker TB, et al. Treating Tobacco Use and Dependence: 2008 Update. Rockville, MD: U.S. Department of Health and Human Services. Public Health Service; 2008.
- [Background] http://www.pewinternet.org/. Accessed January 12, 2010, 2010.
- [Background] Birmingham-Hoover Metropolitan area. Sterling's BestPlaces [http://www.bestplaces.net/Metro/Birmingham-Hoover-Alabama.aspx#. Accessed January 10, 2010.
- [Background] Wolfenden L, Campbell E, Wiggers J, Walsh RA, Bailey LJ. Helping hospital patients quit: what the evidence supports and what guidelines recommend. Prev Med. 2008 Apr;46(4):346-57. doi: 10.1016/j.ypmed.2007.12.003. Epub 2007 Dec 8. PMID 18207229
- [Background] SRNT Subcommittee on Biochemical Verification. Biochemical verification of tobacco use and cessation. Nicotine Tob Res. 2002 May;4(2):149-59. doi: 10.1080/14622200210123581. No abstract available. PMID 12028847
- [Background] Connor Gorber S, Schofield-Hurwitz S, Hardt J, Levasseur G, Tremblay M. The accuracy of self-reported smoking: a systematic review of the relationship between self-reported and cotinine-assessed smoking status. Nicotine Tob Res. 2009 Jan;11(1):12-24. doi: 10.1093/ntr/ntn010. Epub 2009 Jan 27. PMID 19246437
- [Background] Gold MR, Siegel JE, Russel LB, Weinstein MC. Cost-effectiveness in Health and Medicine. New York: Oxford University Press; 1996.
- [Background] Briggs AH, O'Brien BJ, Blackhouse G. Thinking outside the box: recent advances in the analysis and presentation of uncertainty in cost-effectiveness studies. Annu Rev Public Health. 2002;23:377-401. doi: 10.1146/annurev.publhealth.23.100901.140534. Epub 2001 Oct 25. PMID 11910068
- [Background] Doshi JA, Glick HA, Polsky D. Analyses of cost data in economic evaluations conducted alongside randomized controlled trials. Value Health. 2006 Sep-Oct;9(5):334-40. doi: 10.1111/j.1524-4733.2006.00122.x. PMID 16961551
- [Background] Barber JA, Thompson SG. Analysis of cost data in randomized trials: an application of the non-parametric bootstrap. Stat Med. 2000 Dec 15;19(23):3219-36. doi: 10.1002/1097-0258(20001215)19:233.0.co;2-p. PMID 11113956
- [Derived] Triant VA, Grossman E, Rigotti NA, Ramachandran R, Regan S, Sherman SE, Richter KP, Tindle HA, Harrington KF. Impact of Smoking Cessation Interventions Initiated During Hospitalization Among HIV-Infected Smokers. Nicotine Tob Res. 2020 Jun 12;22(7):1170-1177. doi: 10.1093/ntr/ntz168. PMID 31687769
- [Derived] Kathleen F H, Young-Il K, Meifang C, Rekha R, Maria P, Rajani S S, Thomas K H, William C B. Web-Based Intervention for Transitioning Smokers From Inpatient to Outpatient Care: An RCT. Am J Prev Med. 2016 Oct;51(4):620-9. doi: 10.1016/j.amepre.2016.04.008. PMID 27647062
- [Derived] Duffy SA, Cummins SE, Fellows JL, Harrington KF, Kirby C, Rogers E, Scheuermann TS, Tindle HA, Waltje AH; Consortium of Hospitals Advancing Research on Tobacco (CHART). Fidelity monitoring across the seven studies in the Consortium of Hospitals Advancing Research on Tobacco (CHART). Tob Induc Dis. 2015 Sep 3;13(1):29. doi: 10.1186/s12971-015-0056-5. eCollection 2015. PMID 26336372
- [Derived] Harrington KF, McDougal JA, Pisu M, Zhang B, Sadasivam RS, Houston TK, Bailey WC; CHART Collaborative Group. Web-based smoking cessation intervention that transitions from inpatient to outpatient: study protocol for a randomized controlled trial. Trials. 2012 Aug 1;13:123. doi: 10.1186/1745-6215-13-123. PMID 22852802